CLINICAL TRIAL: NCT00486577
Title: Chronic Electrical Stimulation of the Auditory Cortex for Intractable Tinnitus
Acronym: ACOUSCO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Promo 2005
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Hearing Disorders; Hearing Loss; Hyperacusis; Tinnitus
Keywords: Hearing Disorders, Hearing Loss, Hyperacusis, Tinnitus, chronic cortical stimulation, functional magnetic resonance imaging
MeSH Terms: conditions — Hearing Disorders; Hearing Loss; Hyperacusis; Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: significant chronic primary auditory cortex stimulation during the first two weeks
- 2 (Experimental)
  Interventions: Procedure: non significant chronic primary auditory cortex stimulation during the first two weeks

INTERVENTIONS:
Procedure: significant chronic primary auditory cortex stimulation during the first two weeks — significant chronic primary auditory cortex stimulation during the first two weeks of the follow up than wash out period followed by two weeks of non significant stimulation
  Arms: 1
Procedure: non significant chronic primary auditory cortex stimulation during the first two weeks — non significant stimulation during the first two weeks of the follow up than wash out period followed by two weeks of significant chronic primary auditory cortex stimulation
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether chronic electrical stimulation of the primary auditory cortex is effective in the treatment of chronic, severe and intractable tinnitus

DETAILED DESCRIPTION:
Severe and chronic tinnitus - the perception of sound in one or both ears or in the head when non-external sound is present - can be disabling and difficult to treat. Physiopathology of tinnitus can be considered as similar to neuropathic pain. Neuropathic and central pain are treated since ten years by chronic electrical motor cortex stimulation. The hypothesis of this study is that it will be possible to treat severe tinnitus by this stimulation as neuropathic pains are treated by motor cortical stimulation.

* Principal Objective : to evaluate the efficacy of chronic electrical stimulation of the auditory cortex for intractable tinnitus
* Secondary Objective : to evaluate the tolerability and the safety of chronic electrical stimulation of the auditory cortex for intractable tinnitus
* Study design : randomized, cross over, double blind, study to evaluate the efficacy of the chronic electrical stimulation versus sham in severe and chronic tinnitus
* Inclusion criteria :

Patient >18 years of age and < 70 years of age Permanent and chronic tinnitus during more than 2 years. A score over 19 at the STI (Quality of life index for tinnitus) Unilateral tinnitus

• Exclusion criteria : Deaf person Surgical or anesthetic contraindication History of psychiatric disorder or suicide Epilepsia

• Number of subjects : 10

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years of age and < 70 years of age
* Permanent and chronic tinnitus during more than 2 years
* A score over 19 at the STI (Quality of life index)

Exclusion Criteria:

* Deaf person
* Surgical or anesthetic contraindication
* History of psychiatric disorder or suicide
* Epilepsia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
intensity of the tinnitus. The cut off efficacy is 35% improvement on the STI score | 6 months

SECONDARY OUTCOMES:
Tinnitus Handicap Questionnaire Multiple Activity Scale for Hyperacusis questionnaires for assessment of the patients and treatment outcome of tinnitus hyperacusis and loss of hearing subjective global improvement scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Cuny, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- University Hospital of Bordeaux - Pellegrin, Bordeaux, Bordeaux, France

REFERENCES:
- [Derived] Engelhardt J, Dauman R, Arne P, Allard M, Dauman N, Branchard O, Perez P, Germain C, Caire F, Bonnard D, Cuny E. Effect of chronic cortical stimulation on chronic severe tinnitus: a prospective randomized double-blind cross-over trial and long-term follow up. Brain Stimul. 2014 Sep-Oct;7(5):694-700. doi: 10.1016/j.brs.2014.05.008. Epub 2014 Jun 4. PMID 25017670